CLINICAL TRIAL: NCT00355901
Title: An Observational Follow-up Study for Subjects Receiving Salvage Therapy After Previous Treatment in a Visilizumab Study for Intravenous Steroid-Refractory Ulcerative Colitis
Status: Terminated | Type: Observational
Sponsor: PDL BioPharma, Inc. (Industry)
Organization: Facet Biotech (Industry)
Other Study IDs: 291-420
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Colitis; Steroid-Refractory; Visilizumab; Intravenous Steroid-Refractory Ulcerative Colitis (IVSR-UC)
MeSH Terms: conditions — Colitis, Ulcerative; Colitis | interventions — visilizumab

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Visilizumab (Nuvion®; HuM291)

SUMMARY:
To assess the effects of visilizumab on the safety of subsequent salvage therapies in subjects who experienced disease progression in a previous visilizumab study and subsequently received salvage therapy.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in a visilizumab study of IVSR-UC.
* Disease progression while enrolled in a previous visilizumab study, and subsequent treatment with salvage therapy.

Exclusion Criteria:

* Unable to understand the purpose and risks of the study, or unwilling or unable to provide a signed and dated informed consent.
* For U.S. sites, unwilling or unable to provide authorization to use protected health information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-09; Study Completion 2012-11

CONTACTS AND LOCATIONS:
Locations (39):
- United States (14):
  - San Francisco, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Louisville, Kentucky
  - Worcester, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - Manhasset, New York
  - Mineola, New York
  - New York, New York
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Charleston, South Carolina
  - Salt Lake City, Utah
- Australia (4):
  - Bedford Park, South Australia
  - Box Hill, Victoria
  - Fremantle
  - Liverpool
- Vienna, Austria
- Belgium (3):
  - Ghent
  - Leuven
  - Roeselare
- Canada (2):
  - Winnipeg, Manitoba
  - Hamilton, Ontario
- Czechia (2):
  - Brno
  - Prague
- France (3):
  - Amiens
  - Lille
  - Paris
- Freiburg im Breisgau, Germany
- Hungary (3):
  - Béri Balogh Adám
  - Vác
  - Vásvari Pál
- Dublin, Ireland
- Bologna, Italy
- Amsterdam, Netherlands
- Norway (2):
  - Oslo
  - Tromsø
- Kharkiv, Ukraine